CLINICAL TRIAL: NCT06983613
Title: New Onset of Atrial Fibrillation After Percutaneous Patent Foramen Ovale Closure - Na Homolce Hospital
Brief Title: New Onset of Arrhythmia After Patent Foramen Ovale (PFO) Closure
Status: Recruiting | Type: Observational
Sponsor: Na Homolce Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Nemocnice Na Homolce IG250501
Record Dates: First submitted 2025-03-07; First posted 2025-05-21 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-04

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Embolic stroke of undetermined source (ESUS) accounts for approximately 25% of all ischemic strokes, with patent foramen ovale (PFO) considered a major mechanism behind ESUS. When specific anatomic criteria are met, transcatheter PFO occlusion is regarded as the gold standard for secondary stroke prevention.

However, previous studies have shown that percutaneous PFO closure may increase the risk of new-onset atrial fibrillation and atrial flutter (AF), arrhythmias that elevate the risk of embolic stroke. This raises concerns about performing PFO closure. Indeed, the most common clinically significant complication after catheter-based PFO closure is AF. Available data indicates that AF typically occurs in the early period following occluder implantation, with peak incidence around the 14th day post-closure, followed by a decline after the 45th day. Although AF is considered the most frequent adverse complication after percutaneous PFO occlusion, its incidence remains relatively low, ranging from 3% to 7.4%, depending on the method used for arrhythmia screening, though this remains unclear.

In this study, investigators will prospectively monitor patients who have experienced ESUS and are indicated for PFO closure. They will be screened for the occurrence of AF following percutaneous PFO closure using a 3-week ECG Holter monitor (from day 7 to day 28 post-closure) and again 1 week (one year post-closure) after the procedure. The study aims to determine the true incidence of new-onset AF following catheter-based PFO occlusion and to identify the risk factors associated with its development.

ELIGIBILITY:
Inclusion Criteria:

* Indication for percutaneous closure of patent foramen ovale due to stroke, confirmed through an interdisciplinary meeting between cardiologists and neurologists, in accordance with current guidelines.
* Age > 18 years.
* Written informed consent.

Exclusion Criteria:

* Patients with a known history of atrial fibrillation, atrial flutter, or atrial tachycardia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include patients who have experienced ischemic stroke attributed to patent foramen ovale and for whom percutaneous closure has been recommended.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-01-15 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
New onset of atrial fibrillation after percutaneous patent foramen ovale closure - Na Homolce Hospital | 2025-2028
  The primary endpoint - Number of participants with at least 1 episode of atrial arrythmia (atrial fibrillation, atrial flutter, atrial tachycardia), defined as any episode of atrial fibrillation, atrial flutter, or atrial tachycardia lasting ≥ 30 seconds recorded on external cardiac monitor (ECG-Holter) during follow-up.

SECONDARY OUTCOMES:
Time to first episode of atrial arrythmia (atrial fibrillation, atrial flutter, atrial tachycardia) . | 2025-2028
Number of participants with new stroke or transient ischemic attack during follow up. | 2025-2028
Risk factor at baseline. | 2025-2028
  Age - in years (at time of the procedure).
Risk factor at baseline. | 2025-2028
  Weight - in kilograms
Risk factor at baseline. | 2025-2028
  Height - in centimetres
Risk factor at baseline. | 2025-2028
  Body mass index (BMI) - in kg/m2
Risk factor at baseline. | 2025-2028
  Sex - male/female
Risk factor at baseline. | 2025-2028
  CHA₂DS₂-VASc Score for Atrial Fibrillation Stroke Risk
Risk factor at baseline. | 2025-2028
  Risk of Paradoxical Embolism (RoPE) Score - - in points (0-10)
Risk factor at baseline. | 2025-2028
  Number of participants with atrial hypertension
Risk factor at baseline. | 2025-2028
  Number of participants with Diabetes mellitus
Risk factor at baseline. | 2025-2028
  Number of participants with antidiabetic oral drugs
Risk factor at baseline. | 2025-2028
  Number of participants taking insulin
Risk factor at baseline. | 2025-2028
  Number of participants with hypercholesterolemia
Risk factor at baseline. | 2025-2028
  Number of participants actively smoking
Risk factor at baseline. | 2025-2028
  Number of participants formerly smoking
Risk factor at baseline. | 2025-2028
  Number of participants with peripheral embolism
Risk factor at baseline. | 2025-2028
  Number of participants with deep vein thrombosis
Risk factor at baseline. | 2025-2028
  Number of participants with coronary artery disease
Risk factor at baseline. | 2025-2028
  Left Atrial Volume Index in echocardiography - ml/m2
Risk factor at baseline. | 2025-2028
  Right Atrial Volume Index in echocardiography - ml/m2 or right atrial width/lenght in apical 4 chamber view in mm
Risk factor at baseline. | 2025-2028
  Left ventricle ejection fraction in %
Risk factor at baseline. | 2025-2028
  Left ventricle end-diastolic diameter - in mm
Risk factor at baseline. | 2025-2028
  Number of participants with presence of atrial septal aneurysm (assessed on preclosure echocardiography) defined as a septum mobility ≥10 mm from midline
Risk factor at baseline. | 2025-2028
  Presence of right to left shunt on pre-closure echocardiography - Small shunt referred to the appearance of 3 to 10 microbubbles, mild shunt referred to the appearance of 11 to 20 microbubbles, and severe shunt referred to the appearance of >20 microbubbles in the left atrium within 3 cardiac cycles after opacification of the right atrium
Risk factor at baseline. | 2025-2028
  Length of patent foramen ovale (PFO) canal - measured on transoesophageal echocardiography during the procedure in millimetres
Risk factor at baseline. | 2025-2028
  Height of patent foramen ovale (PFO) canal - measured on transoesophageal echocardiography during the procedure in millimetres, defined as the distance between the septum primum and septum secundum at maximum opening
Risk factor at baseline. | 2025-2028
  Invasive pressure measurement in right and left atrium - during the patent foramen ovale (PFO) closure procedure in mmHg
Risk factor at baseline. | 2025-2028
  Type and size of occluder

CONTACTS AND LOCATIONS:
Locations (1):
- Nemocnice na Homolce, Prague, Czechia